CLINICAL TRIAL: NCT06362226
Title: Optimizing Ocular Outcomes: A Dual-armed Study for Periorbital Burn Management
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20029491
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Periorbital Burns
MeSH Terms: interventions — Steroids; Anti-Bacterial Agents; Maxitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A: 5-FU/Kenalog (Experimental)
  Interventions: Drug: 5-FU/Kenalog
- Group B: Steroid/Antibiotic (Experimental)
  Interventions: Drug: Steroid/Antibiotic (Maxitrol)

INTERVENTIONS:
Drug: Steroid/Antibiotic (Maxitrol) — Group one subjects receive topical maxitrol ophthalmic ointment twice daily for two weeks
  Arms: Group B: Steroid/Antibiotic
Drug: 5-FU/Kenalog — Group two undergoes treatment with a subcutaneous injection of a 5-fluorouracil (5-FU) and Kenalog (triamcinolone) combination (80/20 ratio, 0.3-0.5 mL per session) administered in four sessions, spaced two weeks apart, starting within 48 hours of hospital presentation
  Arms: Group A: 5-FU/Kenalog

SUMMARY:
The purpose of this study is to evaluate the effectiveness in using subcutaneous 5-FU/Kenalog & topical Maxitrol Ophthalmic ointment as different therapeutic adjuncts in the prevention of pathologic remodeling after periorbital burns.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age greater than or equal to 18 years at the time of signing informed consent
* Mechanism of Injury including explosion, thermal, electrical
* Clinical diagnosis of periorbital burn wound
* Second degree or less periorbital or lid bur
* No previous surgical treatment for wound management
* Partial Deep thickness Periorbital burn
* Partial Thickness Burn
* Superficial Burn
* Periocular lesions with globe involvement

Exclusion Criteria:

* Recent surgical intervention for wound
* Full Thickness and or "Third degree Burns"
* Imprisoned Inmates
* Chemical Burn
* Pregnant women
* Individuals whom are not adults >18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of wound healing time | 12 months
  This outcome is comparing the would healing time between the 2 groups. A shorter would healing time would indicate faster recovery.
Comparison of infection rate | 12 months
  This outcome is comparing the infection rate during treatment. A lower infection rate may indicate which treatment is superior to the other.
Comparison of complication rates | 12 months
  Complication rate is assessed through the occurrence of adverse events. A lower complication rate could indicate improved safety and tolerability over one treatment.

SECONDARY OUTCOMES:
Comparison of pain level | 12 months
  This will be assessed through the standardized pain scale. The scale is from 1-5. 1 being no pain and 5 being excruciating pain. A lower pain score suggests better pain management due to improved healing.
Comparison of quality of life | 12 months
  The use of the burns outcome questionnaire (BOQ) to assess the participant's quality of life throughout the study. This is a 17 question questionnaire with each question scale being from 0 to 4. 0 being not at all and 4 being very much. The scores are then added up for a total score. The range of total scores is from 0-68. A higher score may indicate improved well-being with a specific treatment.
Comparison of cosmetic outcome through the Vancouver scar scale (VSS) | 12 months
  Variables in the VSS include pigmentation, vascularity, pliability and height. The range for the total score is 0-13. A lower VSS scores suggest better scar appearance as well as quality.
Comparison of cosmetic outcome through the Patient Observer Scar Assessment Scale (POSAS) | 12 months
  Variables in the POSAS include color, thickness, relief, pliability, surface area and overall opinion. The range for the total score is 11-44. Lower POSAS scores indicate improved scar aesthetics.

CONTACTS AND LOCATIONS:
Overall Officials: Nikisha Richards, MD, FACS, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No